CLINICAL TRIAL: NCT00722423
Title: An Integrated Care Model for Improving HCV Patient Outcomes
Brief Title: An Integrated Care Model for Improving Hepatitis C Virus Patient Outcomes
Acronym: HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-101
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; integrated care; alpha interferon; mental health
MeSH Terms: conditions — Hepatitis C; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Care Model (Experimental): Integrated Care
  Interventions: Behavioral: Integrated care model
- Usual Care Model (Experimental): Usual Care
  Interventions: Behavioral: Usual Care Model

INTERVENTIONS:
Behavioral: Integrated care model — The integrated care intervention follows a manualized protocol consisting of a series of brief intervention tailored to the patients' main barriers to treatment along with a case management approach in which the integrated care mental health provider actively tracks each patients progress through the evaluation and treatment process. The integrated care mental health provider can be a clinical nurse specialist, psychologist, or licensed clinical social worker that has experience and training in the provision of psychiatric and SUD interventions. They will receive additional training on the integrated care protocol. Data will be collected at baseline, pre-treatment, and post-treatment intervals.
  Arms: Integrated Care Model
Behavioral: Usual Care Model
  Arms: Usual Care Model

SUMMARY:
This is a prospective randomized controlled trial comparing two different clinic models for patients with hepatitis C. These patients commonly have mental health problems that are barriers to receiving HCV treatment. Patients giving informed consent will be randomized to a usual care HCV clinic vs. a HCV clinic with the addition of an on-site mental health practitioner who will address psychiatric and substance use issues with the goal of enabling patients to undergo effective antiviral therapy. The major outcome of the study is the number of patients in each group who are "cured" with antiviral therapy. Patients in both groups receive current standard of care.

DETAILED DESCRIPTION:
Impact for Veterans: Treatments are available that can often eliminate the hepatitis C virus (HCV) in infected veterans, resulting in increased life expectancy and quality of life. However, many veterans do not get treated or fail treatment because of a variety of factors. Using a new protocol-based model of care that centers around integrating psychiatric care and case management into VA HCV clinics, it may be possible to increase treatment rates, improve rates of sustained viral response (SVR), and improve health outcomes for veterans with hepatitis C.

Background: The prevalence of hepatitis C virus (HCV) infection among VA patients is 3x higher than in the general population. VA patients with HCV have characteristics linked to increased risk for progression to cirrhosis, such as male sex, high body mass index, tobacco or marijuana use, and a history of heavy alcohol use. Antiviral treatment is the only evidence-based treatment that has been shown to eradicate the HCV virus and reduce the progression of liver fibrosis. However, recent VA data indicate that only about 14% of all HCV-infected VA patients have ever received antiviral therapy. Barriers to receiving antiviral treatment include factors such as pre-existing psychiatric illness, ongoing substance abuse, and other medical co-morbidity. Patients with psychiatric and substance use histories have benefitted from an integrated care approach to HCV care, but a more rigorous study design is required to demonstrate effectiveness.

Primary Objective: To determine the effectiveness of a protocol-based integrated care model for increasing treatment rates and the number of patients with successful antiviral treatment as measured by an increase in percentage of all new HCV patients achieving a sustained virologic response (SVR). We hypothesize that this model will increase the proportion of patients who are fully evaluated for treatment, who initiate treatment, and who complete treatment compared with patients that receive usual care. Secondary Objectives: Assess the effects of an integrated care model on patient involvement in care (appointment attendance) and PROs (substance abuse, depression, anxiety). We hypothesize that veterans managed with the integrated care model will have better attendance at HCV clinic appointments, have improved rates of drug and alcohol abstinence, and fewer psychological symptoms.

Project Methods: The intervention is an integrated clinical care model developed and initially studied at the Minneapolis VA HCV Clinic. The preliminary study found that integrated care resulted in higher treatment rates, higher SVRs, reduced substance use, and improved psychological functioning. Thus, we will use a more rigorous randomized design to study the effectiveness of this intervention at 3 major VA medical centers. All clinic patients will be screened for depression, anxiety, PTSD, or recent SUDs and all patients that screen positive on 1 or more of these measures will be asked to participate. Preliminary data suggest that 85% of HCV clinic patients screen positive on at least one measure. Eligible patients will be randomized to either usual or integrated care at each site. The integrated care intervention follows a manualized protocol consisting of a series of brief intervention tailored to the patients' main barriers to treatment along with a case management approach in which the integrated care mental health provider actively tracks each patients progress through the evaluation and treatment process. The integrated care mental health provider can be a clinical nurse specialist, psychologist, or licensed clinical social worker that has experience and training in the provision of psychiatric and SUD interventions. They will receive additional training on the integrated care protocol. Data will be collected at baseline, pre-treatment, and post-treatment intervals. Clinical data will be obtained from VA medical records by the study coordinator at each site. PROs will be assessed using validated measures. Data will be analyzed using hierarchical linear modeling (HLM) techniques.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C. This is defined as the documentation of the presence of circulating hepatitis C virus by a positive hepatitis C Polymerase Chain Reaction test that is compatible with chronic hepatitis. (Note: no requirement is made for the presence of abnormal liver function tests).
* Patients may be treatment na ve or have received and failed prior antiviral treatment.
* Age 18-75 years.
* Patient must be able to give informed consent.
* All antiviral treatments are administered according to accept standards of care at each site, with appropriate pre-treatment evaluation and on-treatment management and precautions. Liver biopsies are an accepted standard of care for patients with chronic hepatitis C and are obtained as clinically indicated.
* Patients must meet screening criteria for "high risk" for mental health and substance use problems. "High risk HCV patient" is defined as a patient with Beck Depression Inventory-II>10 at screening; active drug use indicated by positive urine screen, self-reported use within 6 months on drug use questionnaire or AUDIT-C test >4, or positive PTSD screen.

Exclusion Criteria:

* Patient unable or unwilling to participate.
* Decompensated liver disease, with active or recent encephalopathy, variceal bleeding, or ascites or CHILD-PUGH class B or C. (Note: patients with a history of decompensated cirrhosis in the past with resolution who are otherwise antiviral treatment candidates in the opinion of the treating physician will be considered candidates.)
* Other significant near term life-threatening diseases (malignancy, unstable angina, severe chronic obstructive pulmonary disease, pulmonary fibrosis, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B Ho, MD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System (154C), Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, Bronx, The Bronx, New York

REFERENCES:
- [Background] Groessl EJ, Sklar M, Cheung RC, Brau N, Ho SB. Increasing antiviral treatment through integrated hepatitis C care: a randomized multicenter trial. Contemp Clin Trials. 2013 Jul;35(2):97-107. doi: 10.1016/j.cct.2013.05.002. Epub 2013 May 10. PMID 23669414
- [Result] Ho SB, Brau N, Cheung R, Liu L, Sanchez C, Sklar M, Phelps TE, Marcus SG, Wasil MM, Tisi A, Huynh L, Robinson SK, Gifford AL, Asch SM, Groessl EJ. Integrated Care Increases Treatment and Improves Outcomes of Patients With Chronic Hepatitis C Virus Infection and Psychiatric Illness or Substance Abuse. Clin Gastroenterol Hepatol. 2015 Nov;13(11):2005-14.e1-3. doi: 10.1016/j.cgh.2015.02.022. Epub 2015 Feb 24. PMID 25724704
- [Derived] Groessl EJ, Liu L, Sklar M, Ho SB. HCV Integrated Care: A Randomized Trial to Increase Treatment Initiation and SVR with Direct Acting Antivirals. Int J Hepatol. 2017;2017:5834182. doi: 10.1155/2017/5834182. Epub 2017 Jul 27. PMID 28819570

RESULTS

PARTICIPANT FLOW:
Groups:
- Integrated Care Model: Patients randomized to Integrated Care (IC) received care delivered according to a manualized protocol by a mid-level mental health provider (MHP) located within each HCV clinic. The protocol included brief psychological interventions and case management provided in collaboration with clinic physicians, nurses, and other mental health providers. The MHP evaluated study participants and provided ongoing interventions designed to treat specific mental health problems. The MHP also facilitated a complete treatment evaluation, encouraged the initiation of antiviral treatment, and served as a regular contact and case manager.
- Usual Care Model: Patients randomized to usual care (UC) received "standard of care" required for HCV patients consistent with current VA treatment guidelines and clinic structures.
Period: Overall Study
Arm/Group | Integrated Care Model | Usual Care Model
Started | 182 | 182
Completed | 182 | 181
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care Model | Usucal Care Model | Total
Number analyzed (Participants) | 182 | 181 | 363
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 181 | 363
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (5.51) | 55.5 (5.79) | 55.4 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 178 | 177 | 355
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 33 | 65
  Not Hispanic or Latino | 69 | 62 | 131
  Unknown or Not Reported | 81 | 86 | 167
Region of Enrollment [Number; unit: participants]
  United States | 182 | 181 | 363

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response Rates
Description: Virus not detected by PCR assay
Time Frame: 12-24 weeks post-treatment
Measure: Number; unit: participants
Groups:
- Usual Care Model: usual care
  Patients receive care as usual in their HCV clinic. This care does not include the co-located mental health provider.
Arm/Group | Integrated Care Model | Usual Care Model
Number analyzed (Participants) | 182 | 181
participants | 29 | 14

2. Secondary Outcome: Antiviral Treatment Rate
Description: Number of patients started antiviral treatment
Time Frame: 12-24 weeks post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Integrated Care Model | Usual Care Model
Number analyzed (Participants) | 182 | 181
percentage of participants | 31.9 | 18.8

ADVERSE EVENTS:
Description: Other not serious adverse events were not collected. Only serious adverse events were collected.
  Specific adverse events were not known for the hospitalization event.
Arm/Group | Integrated Care Model | Usual Care Model
Serious Adverse Events (participants affected / at risk) | 112/182 | 125/181
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Integrated Care Model (N=182) | Usual Care Model (N=181)
Hospitalization Events (General disorders) | 104 | 112 — Subjects with a hospital event
Cardiac Arrest (Cardiac disorders) | 1 | 2 — Led to death
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 — Led to death
Medication Overdose (General disorders) | 1 | 0 — Led to death in IC group
Decompensated Cirrhosis (Gastrointestinal disorders) | 2 | 2 — Led to death
Death (General disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes